CLINICAL TRIAL: NCT06772168
Title: A Multicenter, Randomized, Placebo-controlled, Double-blind, Phase III Trial to Evaluate the Efficacy and Safety of CMG190303 in Patients With Type 2 Diabetes and Dyslipidemia
Brief Title: Evaluate the Efficacy and Safety of CMG190303 in Patients With Type 2 Diabetes and Dyslipidemia
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: CMG Pharmaceutical Co. Ltd (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: CMG1903-104
Record Dates: First submitted 2025-01-08; First posted 2025-01-13 (Actual); Last update posted 2026-01-15 (Actual); Status verified 2025-07

CONDITIONS: Dyslipidemia; Type 2 Diabetes
MeSH Terms: conditions — Dyslipidemias; Diabetes Mellitus, Type 2 | interventions — Rosuvastatin Calcium

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- CMG190303(Dapagliflozin/Rosuvastatin) (Experimental)
  Interventions: Drug: CMG190303(Dapagliflozin/Rosuvastatin)
- Comparator 1: Dapagliflozin/Rosuvastatin placebo (Placebo Comparator)
  Interventions: Drug: Comparator 1: Dapagliflozin/Rosuvastatin placebo
- Comparator 2: Rosuvastatin/Dapagliflozin placebo (Placebo Comparator)
  Interventions: Drug: Rosuvastatin/Dapagliflozin placebo

INTERVENTIONS:
Drug: CMG190303(Dapagliflozin/Rosuvastatin) — 0-8 week: Dapagliflozin 10mg and Rosuvastatin 5mg 8-16 week: Dapagliflozin 10mg and Rosuvastatin 10mg 16-24 week: Dapagliflozin 10mg and Rosuvastatin 20mg
  Arms: CMG190303(Dapagliflozin/Rosuvastatin)
Drug: Comparator 1: Dapagliflozin/Rosuvastatin placebo — 0-24 week: Dapagliflozin 10mg and Rosuvastatin placebo
  Arms: Comparator 1: Dapagliflozin/Rosuvastatin placebo
Drug: Rosuvastatin/Dapagliflozin placebo — 0-8 week: Dapagliflozin placebo and Rosuvastatin 5mg 8-16 week: Dapagliflozin placebo and Rosuvastatin 10mg 16-24 week: Dapagliflozin placebo and Rosuvastatin 20mg
  Arms: Comparator 2: Rosuvastatin/Dapagliflozin placebo

SUMMARY:
The goal of this clinical trial is to learn if drug CMG190303 to treat Type 2 Diabetes and Dyslipidemia in adults. It will also learn about the safety of CMG190303. The main questions it aims to answer are:

-Primary Objectives:

1. To compare the change in HbA1c from baseline to 24 weeks between CMG190303 and Rosuvastatin
2. To compare the change in LDL-C from baseline to 24 weeks between CMG190303 and Dapagliflozin

ELIGIBILITY:
Screening (Visit 1) Inclusion Criteria

1. A male or female adult aged between 19 and 80 in South Korea
2. An individual with type II diabetes and dyslipidemia
3. An individual meeting any of the followings at the time of the screening

   1. Metformin monotherapy: An individual who was on a stable dose of metformin ≥1,000 mg/day as monotherapy for at least 6 weeks prior to screening (for a patient who took a dyslipidemia treatment within 4 weeks from the screening, the patient had to be on a stable dose of metformin ≥1,000 mg/day as monotherapy for at least 2 weeks prior to the screening)
   2. Dual combination therapy: An individual who was on a stable dose of metformin ≥1,000 mg/day for at least 1 week prior to the screening in combination with additional oral diabetes treatment (DPP-4i, TZD, SU)
4. An individual meeting the following criteria for HbA1c at the time of the screening

   1. Metformin monotherapy: An individual with 7.0% ≤ HbA1c ≤ 10.5% whose blood sugar level is not adequately controlled
   2. Dual combination therapy: An individual with 6.5% ≤ HbA1c ≤ 10% whose blood sugar level is not adequately controlled
5. An individual with FPG (Fasting Plasma Glucose) ≤ 270 mg/dL at the time of the screening
6. A patient who did not take a dyslipidemia treatment within 4 weeks from the screening and whose fasting serum lipid test level is 100 mg/dL ≤ LDL-C ≤ 250 mg/dL and TG ≤ 400 mg/dL
7. A patient who took a dyslipidemia treatment within 4 weeks from the screening and was on monotherapy of a statin-class drug as a dyslipidemia treatment for at least 6 weeks prior to the screening (an individual who took omega-3 alone or omega-3 in combination with a statin-class drug is considered to have taken the monotherapy of a statin drug as described here)
8. An individual who voluntarily consented to participating in the clinical study and signed the informed consent form

Randomization (Visit 2) Inclusion Criteria

1. An individual who continuously took metformin ≥1,000 mg/day before the randomization (after the screening visit (Visit 1)) and underwent the wash-out period, TLC and run-in period as described below

   1. An individual who took metformin monotherapy but did not take a dyslipidemia treatment: An individual who underwent the TLC for 2 weeks and the TLC and placebo run-in period at the same time for 2 weeks
   2. An individual who took metformin monotherapy and took a dyslipidemia treatment: An individual who underwent the wash-out period for at least 4 weeks, the TLC for 2 weeks, and the TLC and placebo run-in period at the same time for 2 weeks
   3. An individual who took a dual combination therapy of an oral diabetes treatment other than metformin and did not take a dyslipidemia treatment: An individual who underwent the wash-out period for at least 6 weeks, the TLC for 2 weeks, and the TLC and placebo run-in period at the same time for 2 weeks
   4. An individual who took a dual combination therapy of an oral diabetes treatment other than metformin and took a dyslipidemia treatment: An individual who underwent the wash-out period for at least 6 weeks, the TLC for 2 weeks, and the TLC and placebo run-in period at the same time for 2 weeks
2. An individual with 7.0% ≤ HbA1c ≤ 10.5% based on the central laboratory test on a visit 1-4 (Run-in visit)
3. An individual with FPG (Fasting Plasma Glucose) ≤ 270 mg/dL based on the central laboratory test on a visit 1-4 (Run-in visit)
4. An individual whose fasting serum lipid test level is 100 mg/dL ≤ LDL-C ≤ 250 mg/dL and TG ≤ 400 mg/dL based on the central laboratory test on a visit 1-4 (Run-in visit)
5. An individual with medication compliance of 70% or higher during the run-in period

Screening Visit (Visit 1) Exclusion Criteria

1. A patient with hypersensitivity to the active ingredient (dapagliflozin or rosuvastatin) or any component of the investigational product
2. A pregnant woman, a breastfeeding woman, or a woman of childbearing potential or a man who does not agree to use an appropriate contraceptive method* during the clinical study

   *: a. Implantation of an intrauterine device or intrauterine system, b. Dual barrier method for men or women of childbearing potential (condom and contraceptive vaginal diaphragm, vaginal sponge or cervical cap), c. Sterilization (vasectomy, bilateral tubal ligation, etc.)
3. A patient with the body mass index (BMI) < 15 kg/m2 or > 40 kg/m2
4. An individual with the following medical history or laboratory test abnormality

   1. A patient with type I diabetes or secondary diabetes or severe diabetes complications
   2. A patient with metabolic acidosis such as diabetic ketoacidosis
   3. A patient with acute arterial disease at the time of screening (e.g., a patient with a medical history of unstable angina, myocardial infarction, transient ischemic attack, cerebrovascular disease, coronary artery bypass graft, or coronary intervention within 3 months prior to entry to the study)
   4. A patient with a medical history of severe heart failure (NYHA class III to IV), severe heart valve disease, severe obstructive/hypertrophic myocardial disease, severe obstructive coronary artery disease, abdominal aneurysm, or uncontrolled arrhythmia, that occurred within 24 weeks prior to the screening
   5. A patient with uncontrolled hypertension (systolic blood pressure ≥ 180 mmHg or diastolic blood pressure ≥ 110 mmHg) or hypotension (systolic blood pressure < 90 mmHg or diastolic blood pressure < 60 mmHg)
   6. An individual with uncontrolled thyroid dysfunction (TSH (Thyroid Stimulating Hormone) ≥ 1.5 X ULN, or an inability to maintain a stable TSH level in the opinion of the investigator)
   7. An individual with a medical history of myopathy, including rhabdomyolysis, or whose CK is 2 times or higher the upper limit of normal range of CK
   8. A patient with severe renal impairment (eGFR < 45 mL/min/1.73 m2 for a patient taking metformin at 1,000 mg, or eGFR < 60 mL/min/1.73 m2 for a patient taking metformin at > 1,000 mg) or hepatic impairment (AST or ALT is 2.5 times the upper limit of normal range)
   9. An individual with a past history of drug addiction or alcoholism within 1 year from the screening
   10. An individual with major psychiatric disease: Schizophrenia, mood disorder (depression, bipolar disorder), anxiety disorder, obsessive disorder, eating disorder, personality disorder, etc.
   11. Pancreatitis or pancreatic surgery
   12. Urinary tract infection, reproductive system infection (including fungal infection) or urination disorder (exceptionally, an individual who has no urination disorder symptom due to drug treatment, etc. may be enrolled) within 24 weeks from the screening
   13. An individual with a history of a surgery to treat obesity or a gastrointestinal surgery, or a gastrointestinal disorder that impairs drug absorption
   14. A patient with a genetic problem such as galactose intolerance, Lapp lactase deficiency or glucose-galactose malabsorption
   15. An individual in whom a malignancy occurred within 5 years from the screening (exceptionally, an individual who was assessed to have achieved complete response after treatment and did not experience recurrence within at least 2 years from the screening or, regarding basal cell carcinoma, skin epithelial squamous cell cancer, thyroid cancer or intraepithelial carcinoma in other sites, an individual, even with a medical history of the aforementioned cancer within 5 years, who was successfully treated and did not experience recurrence for at least 3 years, may be enrolled depending on the opinion of the investigator)
5. An individual with a history of administering any of the following drugs within 3 months prior to the screening

   1. Insulin injection (exceptionally, an individual who temporarily (for not longer than 14 days) was administered insulin due to surgery or examination may be included) or GLP-1 analogue
   2. Weight control drugs or, in the opinion of the investigator, drugs that may significantly affect weight control
   3. Cyclosporin
6. An individual who has a history of administering a systemic steroid agent within 2 weeks from the screening and requires administration of a systemic steroid agent during the clinical study
7. An individual who is scheduled to have an examination using an iodine contrast agent, or is contraindicated to use of metformin due to acute and chronic metabolic acidosis, etc.
8. An individual who is expected to use a 7.6.1 prohibited concomitant drug during the clinical study, including the screening (use of any prescription drugs and over-the-counter drugs, including prohibited concomitant drugs, must be discussed with the investigator prior to use)
9. A patient who participated in another clinical study and used/applied another investigational product and medical device within 3 months (exceptionally, a patient who participated in a non-interventional observation study may participate in the present study)
10. A patient otherwise considered ineligible for participation in the clinical study in the opinion of the investigator

Randomization Visit (Visit 2) Exclusion Criteria

1. An individual who is not eligible based on recheck of the inclusion/exclusion criteria at the time of randomization
2. An individual who does not fall under the above condition but is otherwise considered ineligible in the opinion of the investigator

Ages: 19 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 240 (Estimated)
Dates: Start 2024-04-19 (Actual); Primary Completion 2026-11-04 (Estimated); Study Completion 2027-02-01 (Estimated)

PRIMARY OUTCOMES:
To compare the change in HbA1c (%) | From enrollment to the end of treatment at 24 weeks
  from baseline to 24 weeks between the dapagliflozin and rosuvastatin combination group and the rosuvastatin monotherapy group
To compare the percentage change in LDL-C | From enrollment to the end of treatment at 24 weeks
  from baseline to 24 weeks between the dapagliflozin and rosuvastatin combination group and the dapagliflozin monotherapy group

SECONDARY OUTCOMES:
To compare the change in HbA1c (%) | From enrollment to the end of treatment at 24 weeks
  from baseline to 24 weeks between the dapagliflozin and rosuvastatin combination group and the dapagliflozin monotherapy group
The percentage change in LDL-C | From enrollment to the end of treatment at 24 weeks
  from baseline to 8, 16, and 24 weeks after administration of the investigational medicinal product
The proportion of subjects achieving LDL-C target levels by cardiovascular risk category | From enrollment to 8, 16, and 24 weeks
  from baseline to 8, 16, and 24 weeks after administration of the investigational medicinal product
The change in fasting plasma glucose (FPG) (mg/dL) | From enrollment to 8, 16, and 24 weeks
  from baseline to 8, 16, and 24 weeks after administration of the investigational medicinal product
The percentage change in the following lipid parameters | From enrollment to 8, 16, and 24 weeks
  from baseline to 8, 16, and 24 weeks after administration of the investigational medicinal product: Total cholesterol (TC) (mg/dL) Triglyceride (TG) (mg/dL) HDL-C (mg/dL) Non-HDL-C (mg/dL) ApoB (mg/dL), ApoAI (mg/dL), ApoB/ApoAI Ratio
The change in HbA1c (%) | From enrollment to the end of treatment at 24 weeks
  from baseline to 24 weeks in the rosuvastatin monotherapy group

OTHER OUTCOMES:
The proportion of subjects with HbA1c < 6.5% | From enrollment to 8, 16, and 24 weeks
  at 8, 16, and 24 weeks from baseline after administration of the investigational medicinal product
The change in blood pressure (SBP/DBP) (mmHg) | From enrollment to 8, 16, and 24 weeks
  from baseline to 8, 16, and 24 weeks after administration of the investigational medicinal product
The change in body weight (kg) | From enrollment to 8, 16, and 24 weeks
  from baseline to 8, 16, and 24 weeks after administration of the investigational medicinal product
The proportion of subjects who used rescue medication and the associated change in HbA1c (%) from baseline to 24 weeks | From enrollment to 8, 16, and 24 weeks

CONTACTS AND LOCATIONS:
Locations (24):
- South Korea (24):
  - Hallym university sungsim medical center, Anyang
  - Buchon sejong hospital, Buchon
  - Inje university heaundea paik hospital, Busan
  - Soonchunhyang cheonan university hospital, Cheonan
  - Keimyung University Dongsan Medical Center, Daegu
  - Daejeon eulji medical center, eulji university, Daejeon
  - Myongji Hospital, Goyang-si
  - Hanyang University Medical Center, Guri-si
  - Chosun University Hospital, Gwangju
  - Wonkwang university hospital, Iksan
  - Inha university hospital, Inchon
  - Chonbuk National University Hospital, Jeonju
  - Bundang CHA medical center, Seongnam
  - Seoul National University Bundang Hospital, Seongnam
  - Nowon eulji medical center, eulji university, Seoul
  - Korea University ANAM Hospital, Seoul
  - Severance hospital, Seoul
  - Kyung hee university hospital at gangdong, Seoul
  - The Catholic University of Korea, Seoul ST. Mary's Hospital, Seoul
  - Hallym university gangnam medical center, Seoul
  - Korea University Guro Hospital, Seoul
  - Ajou University Hospital, Suwon
  - Wonju serverance christian hospital, Wŏnju
  - Yongin Severance Hospital, Yongin-si

IPD SHARING:
Plan to Share IPD: Undecided